CLINICAL TRIAL: NCT03209414
Title: Frailty Syndrome in Daily Practice of Interventional Cardiology Ward
Acronym: FRAPICA
Status: Recruiting | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Andrzej Tomasik MD PhD FESC, Assistant professor, Medical University of Silesia
Other Study IDs: Protocol ver. 1 08 May 2017
Record Dates: First submitted 2017-06-24; First posted 2017-07-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Frail Elderly Syndrome; Coronary Heart Disease; Acute Coronary Syndrome; Coronary Artery Bypass Grafting; Percutaneous Transluminal Coronary Angioplasty
Keywords: Frailty syndrome; Coronary heart disease; Coronary revascularization; Major adverse cardiovascular events; Arterial stiffness; Applanation tonometry; Lean body mass; ST2 biomarker
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4 ml of blood plasma is frozen at -80 degrees of Celsius. SST2 will be assayed after completion of recruitment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stable coronary artery disease: Patients with stable effort angina wil be enrolled. Based on coronary angiography, heart team will decide on medical, percutaneous angioplasty, or bypass grafting.
- Unstable coronary artery disease: Patients with unstable angina wil be enrolled. Based on coronary angiography, heart team will decide on medical, percutaneous angioplasty, or bypass grafting.
- Non-ST elevation myocardial infarction: Patients with non-ST elevation myocardial infarction wil be enrolled. Based on coronary angiography, heart team will decide on medical, percutaneous angioplasty, or bypass grafting.
- ST-elevation myocardial infarction: Patients with ST elevation myocardial infarction wil be enrolled. In majority of patients primary percutaneous coronary intervention will be performed. Based on coronary angiography, heart team will decide on further medical treatment, percutaneous angioplasty, or bypass grafting.

SUMMARY:
The impact of frailty on immediate and long term outcomes of invasive treatment of coronary artery disease is not fully characterized. The assessment of frailty may help physicians in the selection of best treatment option and in the timing and modality of the follow-up. The FRAilty syndrome in daily Practice of Interventional CArdiology ward (FRAPICA) study is designed with the aim to validate the use of the Fried frailty scale and instrumental activities of daily living scale (IADL) as prognostic tools in patients admitted to hospital for symptomatic coronary artery disease, either stable, unstable, or acute coronary syndrome (ACS).

The FRAPICA study is a single center prospective study enrolling patients aged ≥65 years. The aims are (1) to describe Fried frailty scale and IADL scale distribution before hospital discharge and (2) to investigate the prognostic role of Fried frailty and IADL scores. The outcomes are: (1) results of invasive treatment, (2) its complications (periinterventional MI, contrast-induced nephropathy, blood loss), (3) three-year all-cause mortality, cardiovascular mortality, stroke, myocardial infarction, reintervention, heart failure, hospital readmission for any cause, and a composite of the above mentioned. Ancillary analyses will be focused on different clinical presentations, different tools to assess frailty and risk stratification.

The FRAPICA program will fill critical gaps in the understanding of the relation between frailty, cardiovascular disease, interventional procedures and outcome. It will enable more personalized risk assessment and identification of new targets for interventions.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65
* symptomatic coronary artery disease A) stable B) unstable C) NSTEMI D) STEMI
* written, informed consent

Exclusion Criteria:

* lack of consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The investigators assume to enroll consecutive 1000 patients with symptomatic coronary artery disease admitted to 2nd Dept. of Cardiology in Zabrze, Medical University of Silesia for coronary angiography or interventional treatment of the disease. Patients of both sexes aged ≥ 65 years are eligible. An information on study rationale, objectives, and methodology is presented to patients and written, informed consent is required to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Predischarge distribution of frailty syndrome according to Fried phenotype frailty scale | Up to hospital discharge, on average day 4
  Patients will be assessed with Fried frailty scale
Predischarge distribution of frailty syndrome according to instrumental activities of daily living scale | Up to hospital discharge, on average day 4
  Patients will be assessed with instrumental activities of daily living scale

SECONDARY OUTCOMES:
Results of interventional treatment | Up to hospital discharge, on average day 4
  Number of patients with successful revascularization
Incidence of periprocedural infarction | Up to hospital discharge, on average day 4
  Number of patients with periprocedural infarction
Incidence of contrast induced nephropathy | Up to hospital discharge, on average day 4
  Number of patients with contrast induced nephropathy
Incidence of bleeding | Up to hospital discharge, on average day 4
  Number of patients with bleeding
Major cardiovascular events | 36 months
  Number of cardiovascular deaths in long term follow-up
Major cardiovascular events | 36 months
  Number of all-cause deaths in long term follow-up
Major cardiovascular events | 36 months
  Number of patients with reinfarction in long term follow-up
Major cardiovascular events | 36 months
  Number of patients with target lesion revascularization in long term follow-up
Major cardiovascular events | 36 months
  Number of patients with stroke in long term follow-up
Major cardiovascular events | 36 months
  Number of patients with new onset heart failure in long term follow-up
Major cardiovascular events | 36 months
  Number of patients rehospitalized for any cause in long term follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- II Dept. of Cardiology in Zabrze Medical University of Silesia, Zabrze, Upper Silesia, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Woloszyn-Horak E, Salamon R, Chojnacka K, Brzosko A, Bieda L, Standera J, Ploszaj K, Stepien E, Nowalany-Kozielska E, Tomasik A. Frailty syndrome in daily practice of interventional cardiology ward-rationale and design of the FRAPICA trial: A STROBE-compliant prospective observational study. Medicine (Baltimore). 2020 Jan;99(5):e18935. doi: 10.1097/MD.0000000000018935. PMID 32000408